CLINICAL TRIAL: NCT06924723
Title: Effect of Standardized Lacrimal Sac Massage Compared With Probing for Congenital Lacrimal Duct Obstruction: a Non-inferiority, Randomized Clinical Trial
Brief Title: Effect of Standardized Lacrimal Sac Massage Compared With Probing for Congenital Lacrimal Duct Obstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025KYPJ036
Record Dates: First submitted 2025-04-05; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Nasolacrimal Duct Obstruction
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control subjects (Active Comparator)
  Interventions: Procedure: tear duct probing
- experimental group (Experimental)
  Interventions: Procedure: Lacrimal sac massage

INTERVENTIONS:
Procedure: tear duct probing — In-office tear duct exploratory surgery was performed on the study participants, and the children were closely monitored for healing after the procedure.
  The children were closely monitored for healing afterward, and the patients were also examined at 1 week, 1 month, and 2 months after the start of treatment.
  Arms: control subjects
Procedure: Lacrimal sac massage — At the time of the visit, the patient's parents (one of them) were given Standardized tear duct massage (Crigler massage)Teaching and hands-on practice were performed, with the researcher confirming the standardization of movements.Subsequent massages were performed by the family member who received the training, and the child's family swiped the card to access the program.completed by the family member of the child, who scanned the code to enter the small program punch card group, according to the standardized process of massage (the frequency of massage was not less than 3 times/day, each time no less than 4 eight beats)And complete the punch card on time (each punch card interval should be greater than 2 hours).(each clock interval should be more than 2 hours).
  Arms: experimental group

SUMMARY:
Congenital nasolacrimal duct obstruction (CNLDO) is a common ophthalmic condition in children, presenting with tearing and pus overflow, with a prevalence of 5%-20% within 1 year of age. Although most cases resolve spontaneously within 1 year of age, some children require treatment. Lacrimal sac massage is a non-invasive, easy and cost-effective conservative treatment that helps to unblock the obstruction by increasing the pressure in the tear duct. Studies have shown that massage has a 93% cure rate in children under 8 months of age. In contrast, tear duct probing is effective but invasive and risky. In recent years, with the development of minimally invasive techniques, lacrimal sac massage has received renewed attention, and studies have shown its efficacy to be comparable to probing. However, there are problems of non-standardized massage timing and techniques in clinical practice, which affects the therapeutic efficacy. This study aims to assess whether the efficacy of standardized dacryocystic massage is not inferior to that of dacryocystorhinostomy through a randomized controlled trial, providing a reference for the treatment of CNLDO.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 3 months to 1 year;
2. Presence of at least one symptom of CNLDO (tear spillage, mucous discharge) in one or both eyes;
3. No surgical treatment for NLD (probing, balloon dilation, tube placement, DCR, etc.);
4. Can cooperate with the examination and subsequent follow-up;
5. Guardians agreed to be enrolled in the study and signed an informed consent form.

Exclusion Criteria:

1. Combination of presenting infections of the conjunctiva and cornea;
2. Combination of other serious ocular surface and intraocular disorders that may affect the therapeutic effect;
3. Congenital malformation syndromes, developmental delays, facial anomalies, facial deformities; history of surgery or injury to the lacrimal duct, history of punctal occlusion, history of lacrimal fistula, history of congenital bulging of the lacrimal sac, history of acute dacryocystitis, history of severe blepharitis, and perinatal abnormalities such as preterm labor, low birth weight, and so on;

Ages: 3 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Treatment success of congenital tear duct obstruction at 3 months of treatment | At 3 months of starting treatment
  Cure rate of congenital lacrimal obstruction at 3 months of treatment: patients with symptoms of lacrimal obstruction (tearing, pus overflow) disappeared are considered cured; lacrimal irrigation patency rate at 3 months of treatment (all lacrimal irrigation fluid goes into the throat, and no reflux is considered to be patency)

SECONDARY OUTCOMES:
Lacrimal flushing patency at 3 months after the start of treatment | at 3 months after the start of treatment
  Whether the tear duct flushing is smooth
Incidence of complications during treatment | at 3 months after the start of treatment
  Counting adverse events over the course of 3 months of treatment
Recurrence of symptoms within 1 month of cure | 1 month after cure
  Observe whether the patient has recurrence of tearing and pus overflow symptoms within 1 month after cure

IPD SHARING:
Plan to Share IPD: No